CLINICAL TRIAL: NCT07075757
Title: In Situ Injection of Anti-angiogenics in Patients With Brain Arteriovenous Malformations Not Eligible for Exclusion Treatment: Phase I Trial
Brief Title: In Situ Injection of Anti-angiogenics in Patients With Brain Arteriovenous Malformations Not Eligible for Exclusion Treatment
Acronym: BLITZ
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP211033; 2023-506991-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Brain Arteriovenous Malformations
Keywords: Brain arteriovenous malformations (bAVM), in situ intra-arterial injection, Bevacizumab
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single in situ intra-arterial injection of bevacizumab (Experimental): 3 Escalating doses of an in situ intra-arterial injection of Bevacizumab (5 mg/kg, 7.5 mg/kg, 10 mg/kg)
  Interventions: Drug: Single in situ intra-arterial injection of bevacizumab

INTERVENTIONS:
Drug: Single in situ intra-arterial injection of bevacizumab — 3 Escalating doses of an in situ intra-arterial injection of Bevacizumab (5 mg/kg, 7.5 mg/kg, 10 mg/kg)

SUMMARY:
Brain arteriovenous malformations (bAVMs) are rare aggressive vascular malformations affecting mostly young and healthy adults. The most frequent revealing condition (in almost 50% of cases) is an intra-cerebral hemorrhage, which is a considerable source of disability and mortality. The only way to prevent a bleeding or a rebleeding is to perform an exclusion treatment (endovascular embolization, microsurgery, stereotactic radiosurgery, or a combination of these techniques). The major drawback of these treatments is the risk of severe complications, which can reach 20%, especially in patients presenting a bAVM with complex angio-architecture (i.e., grade IV to V in the Spetzler Martin grading scale). There is a growing evidence about the strong implication of angiogenesis (mainly mediated by the type A vascular endothelial growth factor [VEGF-A]) on the size and growth of the bAVM and even in the occurrence of bleeding events. Our hypothesis is that an in situ injection of bevacizumab, a monoclonal antibody inhibiting VEGF-A, in patients with bAVM deemed not suitable for exclusion treatment may be safe and help to reduce the nidus volume.

DETAILED DESCRIPTION:
The main objective of this trial is to evaluate the tolerance of 3 escalating doses of an in situ intra-arterial injection of bevacizumab in patients with a brain arteriovenous malformation (bAVM) considered non-suitable for an exclusion treatment to determine the Maximum Tolerated Dose (MTD) using the Dose-Limiting Toxicity rate (DLT) at 30 days after the injection. The dose limiting toxicity (DLT) is defined as the occurrence within 30 days of the in-situ injection of bevacizumab of one of the following events: Symptomatic venous/arterial thromboembolic events (symptomatic pulmonary embolism, symptomatic deep venous thrombosis, symptomatic ischemic stroke related to an arterial occlusion); Severe cytopenia defined as follows: Anemia defined as hemoglobin (Hb) level less than 8.0 g/dL (grade ≥ III, according to the CTCAE v5.0, 2017) Thrombocytopenia < 50 G/L (grade ≥ III, according to the CTCAE v5.0, 2017), Neutropenia < 1000/μL (grade ≥ IV according to the CTCAE v5.0, 2017); hypertension grade ≥ III (CTCAE v5.0, 2017); symptomatic intracranial hemorrhage resulting in transcient or permanent neurological deficit; any bleeding requiring transfusion; leukoencephalopathy grade ≥ III (CTCAE v5.0, 2017); Onset of intractable seizures ≥ Grade III (CTCAE v5.0, 2017); thrombo-embolic complication during the endovascular procedure leading to permanent deficit or to death; Intracranial arterial perforation with the microcatheter or the microguide wire during the endovascular procedure resulting in severe symptomatic hemorrhage (disability or death); any other serious adverse reaction (any untoward medical occurrence in a subject, to whom the medicinal product is administered, and which have a causal relationship with this treatment) resulting in any disability or death.

The secondary objectives and endpoints are to evaluate 1) the tolerance of 3 escalating doses of an in situ intra-arterial injection of bevacizumab in patients with a bAVM considered non-suitable for an exclusion treatment up to 12 months of follow-up; 2) To evaluate the efficacy of an in situ intra-arterial injection of bevacizumab in patients with a bAVM considered non-suitable for an exclusion treatment in terms of :Nidus volume size reduction at 6 and 12 months, Occurrence of cerebral bleeding events up to 12 months, Occurrence of seizures up to 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and < 65 years at the time of inclusion
2. bAVM (i.e.: located in the brain, brain stem or cerebellum)
3. Spetzler-Martin grade IV - V on a brain MRI performed less than 2 months before inclusion
4. History of rupture and/or with intractable symptoms related to the bAVM (i.e.: intractable seizure, steal phenomenon, compressive symptoms)
5. bAVM deemed unsuitable for exclusion invasive treatment
6. Adequate bone marrow function at inclusion :

   * Hemoglobin (Hb) levels more than 13.5 g/dL in males and Hb levels more than 12.5 g/dL in females.
   * Platelet count ≥ 150 G/L
   * Leukocytes count ≥ 3000/μL
   * Neutrophils count ≥ 1500/μL
7. Normal liver function (alanine transaminase [ALT] < 56 UI/L and aspartate aminotransferase [AST] < 40 UI/L) at inclusion
8. Normal renal function (creatinine clearance ≥ 30 ml/min calculated with the Cockcroft-Gault formula) at inclusion
9. Complete COVID-19 vaccinal scheme, according to the French recommendations
10. Affiliation to French Healthcare system (AME excluded)
11. Signed informed consent

Exclusion Criteria:

1. Diffuse bAVM (like proliferative angiopathy) that cannot be assessed in terms of volume by cross-sectional imaging on MRI
2. Inability/contraindication to undergo MRI (Pacemaker, iron metallic items, cochlear implants, claustrophobia)
3. Coagulation disorders (prothrombin time < 50% or Platelet count < 150 G/L)
4. Any congenital predisposition to coagulation disorder
5. Any disease requiring full anticoagulation
6. History of cancer, except baso-cellular carcinoma
7. Congestive cardiac failure
8. Pre-existing coronary disease
9. Unstable medical or psychiatric illness
10. Any history of clinically significant thrombotic episode within the last 6 months
11. Any history of atrial fibrillation
12. Proteinuria (albumin excretion rate > 30 mg/day)
13. Blood hypertension grade ≥ II (CTACE v5.0, 2017)
14. Past history of a gastro-intestinal fistula
15. Past history of a vaginal fistula
16. Past history of open surgery within the last 28 days
17. Infectious syndrome within the last month
18. Any other contra-indication to bevacizumab administration
19. Any contra-indication to general anesthesia
20. Pregnancy or lactating woman
21. Woman without efficacy contraception (combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinence) all along study participation, and until 6 months after the bevacizumab administration, for woman of childbearing potential
22. Seropositivity for HIV, HCV or HBV
23. Severe and proven allergy to iodinated contrast material or Gadolinium
24. Participation in another interventional clinical trial evaluating a health product or any randomized clinical trial
25. Patients under legal protection (tutorship or curatorship) and patient deprived of freedom

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Days 0 (day of the injection) to day 30
  Dose limiting toxicity defined as the occurrence within 30 days of the in situ injection of bevacizumab of one of the following events:
  * Symptomatic venous/arterial thromboembolic events : pulmonary embolism, deep venous thrombosis, ischemic stroke, related to an arterial occlusion
  * Severe cytopenia defined as:Anemia defined as hemoglobin level less than 8.0 g/dL grade ≥ III,Thrombocytopenia < 50 G/L grade ≥ III
    * Neutropenia < 1000/μ L grade ≥ IV
  * Hypertension grade ≥ III
  * Symptomatic intracranial hemorrhage, resulting in transient/permanent neurological deficit
  * Any bleeding requiring transfusion
  * Leukoencephalopathy grade ≥ III
  * Onset of intractable seizures ≥ Grade III
  * Thrombo-embolic complication during the procedure leading to permanent deficit/death
  * Intracranial arterial perforation with the microcatheter/ microguide wire resulting in symptomatic hemorrhage causing any disability/death.
  * Any other serious adverse reaction resulting in any disability or death

SECONDARY OUTCOMES:
Tolerance of escalating doses (3+3) of an in situ intra-arterial injection of bevacizumab | Days 0 (day of the injection) to 12 months
  Incidence and severity of adverse events
Reduction of the nidus volume | at 6 and 12 months
  Nidus volume size reduction as compared with baseline assessment evaluated on MRI (3D GE T1-weighted images with IV Gadolinium)
Occurrence of an intra-cerebral bleeding event | Days 0 (day of the injection) to 12 months
  Occurrence of intra-cerebral bleeding events from the AVM
Occurrence of at least one seizure | Days 0 (day of the injection) to 12 months
  Occurrence of seizures

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Clarençon, Professor, Principal Investigator — Pitié-Salpêtrière Hospital, AP-HP - Neuroradiology department
Locations (5):
- France (5):
  - CHU de Limoges, Hôpital Dupuytren, Limoges
  - CHU de Nancy, Hôpital Central, Nancy
  - APHP, Hôpital Pitié-Salpêtrière, Paris
  - Centre Hospitalier Sainte-Anne, Paris
  - CHU de Rouen, Hôpital Charles-Nicolle, Rouen

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.